CLINICAL TRIAL: NCT00880516
Title: Genetic Factors in Chronic Sinusitis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16749A
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood for DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: Adults with normal sinuses
- case: Adults with chronic sinusitis and positive findings on imaging.

SUMMARY:
The purpose of this study is to learn more about the genetics of chronic sinusitis and identify genes involved in chronic sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Diagnosis of chronic sinusitis or normal sinuses (with verification by imaging.) You must have a recent CT scan showing either normal sinuses or the presence of sinus disease.

Exclusion Criteria:

* Genetic or acquired immunodeficiency
* Ciliary dyskinesia
* Cystic fibrosis
* Autoimmune disease
* Cancer of the sinuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with and without chronic sinusitis
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2009-04-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Association of genetic variation with CRS disease status | Adult age

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Pinto, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States